CLINICAL TRIAL: NCT01413269
Title: Phase 3 Open-labeled Randomized Clinical Study of Comparing Hypofractionated and Conventional Radiotherapy for Breast Cancer Patients After Breast Conservative Surgery
Brief Title: Randomized Study of Hypofractionated and Conventional Fractionation Radiotherapy After Breast Conservative Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, M.D., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-013
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: breast cancer patients; breast conservation surgery; hypofractionated radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypofractionation radiotherapy (Experimental): irradiation to the whole breast to a total dose of 43.5Gy,at 2.9Gy per fraction, 5 fractions a week, followed by tumor bed boost of 8.7Gy, at 2.9Gy per fraction 5 fractions a week.
  Interventions: Radiation: radiotherapy
- conventional fractionation radiotherapy (Active Comparator): irradiation to the whole breast to a total dose of 50Gy,at 2.0Gy per fraction, 5 fractions a week, followed by tumor bed boost of 10Gy, at 2.0Gy per fraction 5 fractions a week.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — one group receives radiation to the whole breast to a total dose of 43.5Gy,at 2.9Gy per fraction, 5 fractions a week, followed by tumor bed boost of 8.7Gy, at 2.9Gy per fraction 5 fractions a week.
  the other group receives radiation to the whole breast to a total dose of 50Gy,at 2.0Gy per fraction, 5 fractions a week, followed by tumor bed boost of 10Gy, at 2.0Gy per fraction 5 fractions a week.

SUMMARY:
Early-stage breast cancer patients treated with breast conservative surgery are enrolled in this study if they meet defined criteria. Patients are randomized into two groups: conventional fractionation radiotherapy and hypofractionated radiotherapy.The hypothesis is that conventional fractionation radiotherapy and hypofractionated radiotherapy have similar efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. KPS>=60
2. histology confirmed invasive breast cancer
3. received breast conservative surgery(wide local excision and axilla dissection, or axillary sentinel node biopsy if sentinel node is negative)
4. surgical margins negative
5. primary tumor ≤5cm in the largest diameter
6. no internal mammary node or supraclavicular node metastases or distant metastasis
7. can tolerate chemotherapy,hormone therapy (if needed) and radiotherapy
8. for patients not need chemotherapy，enrollment date is required no more than 8 weeks from surgery date
9. for patients with chemotherapy first,enrollment date is required no more than 8 weeks from the last date of chemotherapy
10. patients signed written inform consent form

Exclusion Criteria:

1. ductal carcinoma in situ
2. prior neoadjuvant chemotherapy
3. prior breast cancer history
4. bilateral breast cancer
5. pregnant or during lactation
6. prior or concomitant malignant tumor excluded skin cancer(not malignant melanoma) and cervix carcinoma in situ
7. active collagen vascular disease
8. prior neoadjuvant hormone therapy
9. immediate ipsilateral breast reconstruction

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2010-06; Primary Completion 2015-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
in-breast recurrence rate | 5 year
  evidence of ipsilateral breast local recurrence confirmed by histology

SECONDARY OUTCOMES:
regional node recurrence rate | 5 year
  ipsilateral axillary node, internal mammary node and supraclavicular node recurrence confirmed by physical examination, image evaluation or histology.
disease-free survival | 5 year
  locoregional relapse, distant relapse, death
overall survival | 5 year
  any death
acute toxicity | 6 months
  radiation dermatitis and radiation pneumonitis evaluated and graded by CTC3.0 criteria
late complication | 3 -10 year
  breast cosmetic effect, ischemic heart disease, rib fracture, arm edema and shoulder joint dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: ye-xiong Li, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shu-lian Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Beijing hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing

REFERENCES:
- [Derived] Wang SL, Fang H, Hu C, Song YW, Wang WH, Jin J, Liu YP, Ren H, Liu J, Li GF, Du XH, Tang Y, Jing H, Ma YC, Huang Z, Chen B, Tang Y, Li N, Lu NN, Qi SN, Yang Y, Sun GY, Liu XF, Li YX. Hypofractionated Versus Conventional Fractionated Radiotherapy After Breast-Conserving Surgery in the Modern Treatment Era: A Multicenter, Randomized Controlled Trial From China. J Clin Oncol. 2020 Nov 1;38(31):3604-3614. doi: 10.1200/JCO.20.01024. Epub 2020 Aug 11. PMID 32780661